CLINICAL TRIAL: NCT06929780
Title: Prolonged Mechanical Ventilation Following Acute Type A Aortic Dissection Surgery: Risk Factor Analysis, Impact on Clinical Outcomes and Development of Prediction Model
Brief Title: A Prediction Model of Prolonged Mechanical Ventilation Following Acute Type A Aortic Dissection Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Professor, China-Japan Friendship Hospital
Other Study IDs: 2025-zxm-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Acute Type A Aortic Dissection
Keywords: Acute type A aortic dissection; Prolonged mechanical ventilation; mechanical ventilation time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Development cohort: As the development cohort, this cohort retrospectively enrolled approximately 1000 postoperative patients undergoing acute type A aortic dissection (ATAAD) surgery to establish a clinical model for predicting the risk of prolonged mechanical ventilation (PMV) after ATAAD surgery.This cohort will also be utilized to analyze the risk factors for PMV following ATAAD surgery and their impact on clinical outcomes.
- Validation cohort: As the validation cohort, this cohort retrospectively enrolled approximately 400 patients (from January 2024 to December 2024) who underwent ATAAD surgery to validate the predictive performance of the model.

SUMMARY:
The goal of this observational study is to develop and validate a predictive model for prolonged mechanical ventilation (PMV) following acute type A aortic dissection (ATAAD) surgery.

The main questions it aims to answer are:

1. To validate the predictive performance of the model for PMV after ATAAD surgery
2. To assess the proportion of PMV among patients undergoing ATAAD surgery
3. To evaluate the ICU length of stay and operative mortality in patients with PMV following ATAAD surgery

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of acute type A aortic dissection (ATAAD) confirmed by computed tomography angiography and echocardiography;
* Patients who underwent aortic surgery requiring cardiopulmonary bypass (CPB), were admitted to the surgical intensive care unit (SICU), and received mechanical ventilation.

Exclusion Criteria:

* Reintubation;
* Intraoperative death or failure to survive beyond 72 hours postoperatively;
* Pregnancy;
* Severe comorbidities (e.g., lung cancer);
* Missing critical outcome data (e.g., short-term mortality, mechanical ventilation duration, reintubation).

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ATAAD postoperative patients admitted to SICU
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The predictive performance of the model for prolonged mechanical ventilation (PMV) following acute type A aortic dissection (ATAAD) surgery | 72 hours after ATAAD surgery
  The predictive performance of PMV following ATAAD surgery includes its discriminative ability and calibration ablility.
The proportion of patients with PMV | 72 hours after ATAAD surgery
  The proportion of patients with PMV refers to the proportion of patients with PMV among the total included ATAAD postoperative patients. PMV is defined as postoperative mechanical ventilation lasting more than 72 hours

SECONDARY OUTCOMES:
ICU length of stay (ICU-LOS) | From surgery to discharge or death, whichever came first, assessed up to 6 months
  ICU length of stay was defined as the length of time spent in ICU from surgery to discharge or death.
surgery-related mortality | 30 days after ATAAD surgery
  surgery-related mortality encompassed any death occurring during the index hospitalization (even beyond 30 days) or after discharge but before postoperative day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No